CLINICAL TRIAL: NCT02912013
Title: The Efficacy of the Me Mini Device for Hair Removal: A Prospective, Open Label Study With Before-After Design
Brief Title: The Efficacy of the Me Mini Device for Hair Removal
Acronym: OHR2-MeMini
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment rate was not sufficient
Sponsor: Iluminage Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 303-17
Record Dates: First submitted 2016-09-17; First posted 2016-09-23 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Hair Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Me mini (Experimental): Subjects treated with Me mini device
  Interventions: Device: Me Mini

INTERVENTIONS:
Device: Me Mini — Home use hair removal device

SUMMARY:
The Mē Mini is a compact version of the Mē device that was cleared by the FDA for removal of unwanted hair and for permanent hair reduction for all skin colors (Fitzpatrick skin photo-types I-VI) based on a series of multi-site clinical studies.

The purpose of this post-marketing study is to support the claims for removal of unwanted hair and for permanent hair reduction in the compact version of the device.

DETAILED DESCRIPTION:
The purpose of this post-marketing study is to determine the efficacy of the mē mini hair removal device and to compare the extent of hair removal with and without maintenance treatments.

Healthy females, with dark hair in the treatment areas that desire to remove their hair will be enrolled. Subjects will be provided with the device and will be instructed as to the method of usage. The subjects will be expected to self-administer the treatment at the clinic in a "simulated home environment". Subjects will receive 7 "basic treatments" in weekly intervals and 3 additional maintenance treatments on 1 side in 1 month intervals ("Maintenance" vs "No maintenance" side). In the second phase of the study subjects that consented to and completed the first phase will be offered the option to continue with 9 additional maintenance treatments in 1 month intervals.

Follow ups will be conducted at 1, 3, 6, 9, and 12 months after the last basic treatment.

Evaluations will include hair clearance, skin safety, tolerability of the procedure, and subject, satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, between 18 and 65 years of age.
2. Subject has Black or dark brown terminal hairs in the areas to be treated.
3. Terminal hair density requirement of greater than 15 hairs within the hair count site (3x3 cm area) as determined by manual hair count performed by the study investigator.
4. Willing to sign informed consent.
5. Willing to follow the treatment schedule and post treatment follow-up.
6. Willingness to have photographs of the treated area taken that may be used for marketing and educational presentation and/or publications and willing to sign the photo-release form.
7. Willingness to avoid excessive sun exposure two weeks prior to treatments

Exclusion Criteria:

Skin and Hair

1. Subjects with white, red, light brown and/ or blonde hairs in the areas to be treated.
2. A history of keloidal scarring (hypertrophic scars or keloids).
3. Active dermatologic lesion or infection in the treatment site.
4. Subject has permanent tattoos or makeup in the treatment area.
5. Recently tanned in the area to be treated and/or unable or unlikely to refrain from tanning during the study.
6. Subject has disease related to photosensitivity, such as porphyria, polymorphic light eruption, solar urticaria, lupus, etc
7. Subject has a history of herpes outbreak in the area of treatment, unless receiving preventative treatment from physician Other Medical Conditions
8. Pregnant, planning to become pregnant, hormone fluctuations and/or breast feeding during the experiment.
9. Subjects with Diabetes (Type I or II) or other systemic or metabolic condition
10. Subject has an active electrical implant anywhere in the body, such as a pacemaker, an internal defibrillator, insulin pump, incontinence device, etc.
11. Subject suffers from epilepsy.
12. Subject has active cancer, or has a history of skin cancer or any other cancer in the area to be treated, including presence of malignant or pre-malignant pigmented lesions.
13. Subject received radiation therapy or chemotherapy treatments with the past 3 months.
14. Subject has known anticoagulative or thromboembolic condition or is on any form of anticoagulation treatment.
15. Subject has a history of immunosuppressant/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
16. Subject has any other condition which in the physician's opinion would make it unsafe for the subject to be treated.

    Medication/treatments
17. Subject had rotating type tweezer epilator treatment, or waxing within the last 3 months
18. Subject had electrolysis treatment within the last 6 months over the treatment area.
19. Subject had any type of professional intense pulsed light (IPL), laser or RF hair removal in the treatment site within the last 6 months.
20. Subject is taking medication known to induce photosensitivity, including non-steroidal anti-inflammatory agents, tetracyclines, phenothiazines, thiazide diuretics, sulfonylureas, sulfonamides, Dacarbazine(DTIC), fluorouracil, vinblastine, and griseofulvin within 4 weeks of therapy.
21. Subject has been taking Accutane® within 6 months of therapy.
22. Subject has been on steroid regimen during the last three months.
23. Subject is on Gold therapy (for arthritis treatment).
24. Subjects who have participated in any clinical study within the 30 days prior to the first planned treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Hair Clearance at 1 Month Follow up | 3 months after beginning of the study (1 month after completion of 7 weekly treatments that last 2 months)
  Hair clearance = the percent of hair cleared from baseline to endpoint.

SECONDARY OUTCOMES:
Hair Clearance at 3-month (Final) Follow up | 5 months after beginning of the study (3 months after completion of 7 weekly treatments that last 2 months)
  Hair clearance = the percent of hair cleared from baseline to endpoint.
Occurrence of Anticipated Effects on Skin | 1 year and 2 months (throughout the study)
  As with other IPL devices, subjects were informed that they should expect some sense of warmth, tingling, or itching, when the device was applied. This was anticipated to be mild to moderate. Subjects could also expect transient erythema and edema at the treatment site that usually disappears within 24 hours.
Tolerability Level of the Procedure Following Treatments | 1, 3, 7 weeks (basic weekly treatment 1, 3, and 7), and 5, 8, 11, 14 months (maintenance monthly treatment#3, 6, 9, 12)
  Tolerability was rated by the subjects using a 5 point pain scale (no pain, mild pain, moderate pain, severe pain, Intolerable [had to stop treatment]).
Subject Satisfaction | 5, 8, 11, and 14 months
  Gathering information about the subject satisfaction from the hair removal procedure based on 5 point satisfaction scale.

CONTACTS AND LOCATIONS:
Overall Officials: David J Friedman, MD, Principal Investigator — Friedman Laser & Skin Center; Lilach Gavish, PhD, Study Director — HUJI
Locations (1):
- David Friedman, Skin & Laser Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No